CLINICAL TRIAL: NCT03661944
Title: Can Functional Performance Assessments in Overhead Athletes With Shoulder Injury Assess the Ability of Return to Play (RTP)?
Brief Title: Functional Performance Assessments in Overhead Athletes With Shoulder Injury
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807118RINB
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2018-08

CONDITIONS: Sports Physical Therapy; Rehabilitation
Keywords: sports; physical therapy; return to play; overhead athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic group: There is no intervention in this group, only functional assessments and general physical examinations will be done
  Interventions: Diagnostic Test: functional performance test
- Healthy control group: There is no intervention in this group, only functional assessments and general physical examinations will be done
  Interventions: Diagnostic Test: functional performance test

INTERVENTIONS:
Diagnostic Test: functional performance test — Functional performance test is to test the ability of the athletes in functional movements

SUMMARY:
Background & Purpose: Shoulder injuries are commonly seen in overhead athletes due to the mechanism of the repetitive and high velocity movement. While the injury usually cost the lost of time in playing, making the decision of the time to return to play (RTP) is a critical issue that should be standardized and objective. However, current studies showed that the decision making of RTP is so complicated that there's lack of objective measurements especially for upper extremity injuries. So, investigating the usage of convenient and valid tools, functional performance assessments for assessing the ability to RTP is the main objective of this study.

Objective: There are 2 objectives for this study: (1) to investigate the difference between RTP group and non-RTP in overhead athletes with shoulder injury; (2) to investigate the responsiveness of the functional performance assessment in return to play for overhead athletes with shoulder injury. Methods: Overhead athletes with shoulder injury or surgery which leads to temporary leaving to the sport within will be recruited in this study. The shoulder joint range of motion (flexion, extension, external/internal rotation, and abduction), shoulder muscle strength (flexors, abductors and external/internal rotators), patient-reported outcome (KJOC and DASH questionnaire) and functional performance assessments (FMS, YBT-UQ, CKCUEST, USSP and TPUT) will be assessed at 6 months after the athlete was injured or received surgery, and at the time point if the athletes successfully complete at least one formal game or practice game (RTP group). If the athlete doesn't return within 12 months after injury or surgery, the assess will be done at the 12th month after injury or surgery. Significance and Contribution: This study is going to provide an objective measurement value of functional performance assessment in injured overhead athletes, determining whether the strength, endurance or power of the upper extremity is good enough to return to the sport that the athlete played before this injury. The result is also expected to have significant contribution in the area of sports medicine in return to play especially in overhead athletes, which has limited evidence providing specific criteria and objective measurement value previously.

ELIGIBILITY:
Inclusion Criteria:

* overhead athletes diagnosed with shoulder injury within 6 months and can't play the current sports
* accepting the routine rehabilitation
* have the intention to go back to current sports

Exclusion Criteria:

* Other severe orthopedic injuries in upper extremity, lower extremity and spine within 1 year
* has no intention to return to play

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Overhead athletes with shoulder injury
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
FMS | 10 minutes
  functional movement screen
YBTUQ | 10 minutes
  y-balance test upper quarter
USSP | minutes
  unilateral seated shot put test
CKCUEST | 5 minutes
  closed kinetic chain upper extremity stability test
TPUT | 5 minutes
  timed push up test

SECONDARY OUTCOMES:
shoulder range of motion | 10 minutes
  shoulder flexion, extension, abduction, external and internal rotation
shoulder muscle strength | 15 minutes
  shoulder flexion, abduction, external and internal rotation
Disability of Arm, Shoulder and Hand questionnaire | 10 minutes
  patient reported outcome about the functional status of the shoulder The questionnaire is divided into 4 parts, the first part assesses the disability in daily activities, the second part assesses the severity of the symptom, the third and fourth part assesses the disability in working and playing sports or music instruments. The scale is from 1 to 5, which higher points indicates greater disability.
  First and second part will be sum up and get the total score, which higher score indicates greater disability in arm, shoulder or hand region.
  The third and fourth part will be assessed independently, and the score as well as higher scores indicates higher degree of disability in arm, shoulder, and hand region.
KJOC questionnaire | 10 minutes
  patient reported outcome about the functional status of the shoulder This questionnaire contains 10 different items, which are about the performance during overhead sports competition. Each item score ranges from 0 to 10, which higher scores indicate better performance or less change or influence in their performance and each item will be sum up to get the total score. Therefore, the total score ranges from 0 to 100, and the higher the score, the better the functional status they were.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Hung Chao, Principal Investigator — Institution of Physical Therapy, National Taiwan University
Locations (1):
- Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No